CLINICAL TRIAL: NCT05006235
Title: Inhaled Beta-2 Agonist Versus Epinephrine For Treatment of Transient Tachypnea of Newborn
Brief Title: Inhaled Beta-2 Agonist Versus Epinephrine For Treatment of Transient Tachypnea of Newborn (TTN)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ahmed Noaman (Other)
Responsible Party: Sponsor-Investigator, Ahmed Noaman, Lecturer, Mansoura University Children Hospital
Organization: Mansoura University Children Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MansouraUCH0321
Record Dates: First submitted 2021-07-21; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Transient Tachypnea of the Newborn
Keywords: Transient Tachypnea of the Newborn (TTN); epinephrine; salbutamol; respiratory distress; newborn
MeSH Terms: conditions — Transient Tachypnea of the Newborn; Dyspnea | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Salbutamol Group (Active Comparator): included babies who had received nebulized B2 agonist salbutamol (0.15 mg/kg) + 4ml normal saline
  Interventions: Drug: Salbutamol
- Epinephrine Group (Active Comparator): included babies who had received nebulized epinephrine (0, 05 ml/Kg) + 4ml normal saline
  Interventions: Drug: Epinephrine Inhalation Solution
- Saline Group (Placebo Comparator): include babies who had received nebulized 0.9% saline
  Interventions: Drug: Saline Inhalants

INTERVENTIONS:
Drug: Epinephrine Inhalation Solution
  Arms: Epinephrine Group
Drug: Salbutamol
  Arms: Salbutamol Group
Drug: Saline Inhalants
  Arms: Saline Group

SUMMARY:
Inhaled Beta-2 Agonist Versus Epinephrine For Treatment of Transient Tachypnea of Newborn: Randomized controlled trial to assess:

DETAILED DESCRIPTION:
This is a randomized double-blind randomized controlled trial. It had been conducted at the Neonatal Intensive Care Unit (NICU) of Mansoura University Children's Hospital, Egypt Written informed consent had been taken from all parents whose infants were recruited in the study. The ethics committee of the faculty of medicine has approved the study.

ELIGIBILITY:
Inclusion Criteria:

* babies with 35 weeks of gestation or more in the first 6 hours of life diagnosed with TTN according to the criteria of which are:

  * Tachypnea (respiratory rate exceeding 60 breaths/ min) within 6 hours after birth
  * Persistence of tachypnea for at least 12 hours
  * Mild cyanosis, nasal flaring, or retractions.
  * Chest radiograph indicating at least one of the following:
* Prominent central vascular markings
* Widened interlobar fissures
* Symmetrical perihilar congestion
* Hyperaeration is evidenced by flattening and depression of the diaphragmatic domes.

Exclusion Criteria:

* Newborn infants with gestational age < 35 weeks
* Meconium aspiration
* Respiratory distress syndrome
* Pneumonia
* Congenital heart diseases including persistent pulmonary hypertension of the neworn (PPHN)
* Sepsis or suspected sepsis
* Polycythemia
* Newborn infants with congenital malformations and chromosomal anomalies
* Newborn infants with ventilatory support.
* Newborn infants with arrhythmia

Ages: 1 Hour to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 135 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Duration of oxygen support & O2 concentration until Downes' score less than 4 | through study completion, about 1 year

SECONDARY OUTCOMES:
Length of hospital stay until Downes' score less than 4 | through study completion, about 1 year
Type of respiratory support (oxygen delivery and oxygen concentration) | within 12 hours after intervention
Effect of intervention on blood sugar (mg/dl) | within 12 hours after intervention

REFERENCES:
- [Background] Bertrand P, Aranibar H, Castro E, Sanchez I. Efficacy of nebulized epinephrine versus salbutamol in hospitalized infants with bronchiolitis. Pediatr Pulmonol. 2001 Apr;31(4):284-8. doi: 10.1002/ppul.1040. PMID 11288210
- [Background] Clark RH. The epidemiology of respiratory failure in neonates born at an estimated gestational age of 34 weeks or more. J Perinatol. 2005 Apr;25(4):251-7. doi: 10.1038/sj.jp.7211242. PMID 15605071
- [Background] Rawlings JS, Smith FR. Transient tachypnea of the newborn. An analysis of neonatal and obstetric risk factors. Am J Dis Child. 1984 Sep;138(9):869-71. doi: 10.1001/archpedi.1984.02140470067022. PMID 6540983
- [Background] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Plavka R, Saugstad OD, Simeoni U, Speer CP, Vento M, Halliday HL; European Association of Perinatal Medicine. European consensus guidelines on the management of neonatal respiratory distress syndrome in preterm infants--2013 update. Neonatology. 2013;103(4):353-68. doi: 10.1159/000349928. Epub 2013 May 31. PMID 23736015
- [Background] Vollsaeter M, Roksund OD, Eide GE, Markestad T, Halvorsen T. Lung function after preterm birth: development from mid-childhood to adulthood. Thorax. 2013 Aug;68(8):767-76. doi: 10.1136/thoraxjnl-2012-202980. Epub 2013 Jun 7. PMID 23749815
- [Background] Yurdakok M. Transient tachypnea of the newborn: what is new? J Matern Fetal Neonatal Med. 2010 Oct;23 Suppl 3:24-6. doi: 10.3109/14767058.2010.507971. PMID 20807157